CLINICAL TRIAL: NCT01654653
Title: A Phase , Prospective, Randomized, Open-label Study to Compare the Efficacy and Safety of Hypertonic Sodium Lactate Solution Compared With 6% HES Solution in CABG (Coronary Artery Bypass Grafting) Patients
Brief Title: Efficacy and Safety of Hypertonic Sodium Lactate Solution Compared With 6% HES Solution in CABG Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB.05.01.1.4.0.70
Record Dates: First submitted 2012-05-03; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Heart Disease
Keywords: Heart disease; cardiac surgery; CABG; Totilac; Voluven; 6% HES
MeSH Terms: conditions — Coronary Disease; Heart Diseases | interventions — HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HSL(Totilac) (Experimental): Hypertonic Sodium Lactate
  Interventions: Drug: Hypertonic sodium lactate
- 6% HES (Voluven) (Active Comparator): 6% Hydroxyethyl Starch
  Interventions: Drug: 6% Hydroxy Ethyl Starch

INTERVENTIONS:
Drug: Hypertonic sodium lactate — Administered at beginning of surgery as loading dose at 3 mL/kg body weight within 15 minutes. Additional fluid administered if needed and this was was managed similarly in both groups; the types and amount of additional fluid was measured and recorded. Surgery procedure and concomitant medication was managed similarly.
  Other Names: Totilac
  Arms: HSL(Totilac)
Drug: 6% Hydroxy Ethyl Starch — Administered at beginning of surgery as loading dose at 3 mL/kgBW within 15 minutes. Additional fluid given if needed and this was managed similarly in both groups; the types and amount of additional fluid was measured and recorded. Surgery procedure and concomitant medication was managed similarly
  Other Names: Voluven
  Arms: 6% HES (Voluven)

SUMMARY:
The choice of fluid therapy is controversial in cardiac surgery. Numerous studies have shown that colloid is better as compared to crystalloids. Several previous studies have demonstrated that Hypertonic Sodium Lactate (HSL) administration during cardiac surgery shows a promising effect. This study aims to compare hemodynamic effects and fluid balance of HSL with 6% Hydroxy Ethyl Starch (HES).

DETAILED DESCRIPTION:
The primary objectives of this prospective, randomized and open-label study are as follows:

* To evaluate the clinical efficacy of Hypertonic Sodium Lactate (HSL) in comparison with 6% HES to maintain hemodynamic stability in intra CABG patients related to hemodynamic status and Body fluid balance.
* To assess the safety of HSL in intra CABG patients related to defined laboratory parameters clinical adverse events which occur during the trial.

Subjects meeting enrolment criteria will be randomly assigned to HSL or 6%HES treatment groups.

Assessment of comparability will be done by unpaired student t-test or Chi-Square test or by a two-way ANOVA for repeated measures followed by post-hoc analysis when significant difference is found within the two groups.

The hypothesis tested is that HSL is effective in intra CABG surgery patients, requiring less volume with better cardiac index, as compared to 6% HES.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 45-80 years.
* CABG patients with on or off pump procedure.
* Ejection fraction <50%
* Patients who have given their written informed consent.

Exclusion Criteria:

* Combined operations(surgeries)
* Patients with severe arrhythmia (VT, AF rapid response, heart block) and severe hemodynamic imbalance.
* Severe bleeding and/or re-operation.
* Hypernatremia> 155 mmol/L
* Severe liver failure: SGOT and SGPT more than twice normal.
* Severe renal failure: creatinine more than 2 mg%.
* Patients with major diseases such as cancer, etc.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | Assessed from baseline till upto end of surgery(mean duration of surgery was 372.47 ± 122.82 min in HSLgroup vs 380.61 ± 82.08 min in HES group
  • Evaluation of efficacy of Hypertonic Sodium Lactate against 6% HES to maintain hemodynamic stability in intra CABG patients:
  1. Hemodynamic status (CI, MAP, PVR/PVRI, SVR/SVRI, CVP, PAM, PAW, HR).
  2. Body fluid balance (urinary output; total fluid loss including urine and hemorrhage; total fluid infusion including HSL and 6% HES, blood product and other fluids).
Safety | Assessed from baseline till upto end of surgery(mean duration of surgery was 372.47 ± 122.82 min in HSLgroup vs 380.61 ± 82.08 min in HES group
  Assess safety of HSL in intra CABG patients:
  1. Lab parameters: Hb, HCT, Na,K, Cl, Mg, lactate, glucose, and arterial blood gas.
  2. Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Cindy E Boom, PhD, MD, Principal Investigator — National Cardiovascular Center Harapan Kita, Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, Jakarta Special Capital Region, Indonesia